CLINICAL TRIAL: NCT07395960
Title: The Efficacy and Safety of Metformin Intervention in Elderly Overweight or Obesity With Mild Cognitive Impairment by a Single-center, Randomized, Placebo-controlled Interventional Study (Include Elderly Patients With Obesity or Overweight)
Brief Title: The Efficacy and Safety of Metformin Intervention in Elderly Overweight or Obesity With Mild Cognitive Impairment
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Bin Lu, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025K299
Record Dates: First submitted 2025-12-20; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment; Overweight or Obesity; Elderly
MeSH Terms: conditions — Cognitive Dysfunction; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metformin (Experimental): The intervention group was administered metformin sustained-release tablets (taken once daily, 1500mg each time; if intolerable, the dosage was reduced to the maximum tolerated dose).
  Interventions: Drug: Metfomin
- control (No Intervention)

INTERVENTIONS:
Drug: Metfomin — The intervention group is administered metformin sustained-release tablets (taken once daily, 1500mg each time; if intolerable, the dosage was reduced to the maximum tolerated dose).
  Arms: metformin

SUMMARY:
The prevalence of cognitive impairment in elderly obese patients is high, and the burden on families and society is heavy. Early intervention for mild cognitive impairment (MCI) is of great value. Central nervous system insulin resistance plays a role in the pathogenesis of cognitive impairment, and functional magnetic resonance imaging(fMRI) can evaluate cognitive impairment by observing central insulin resistance. Some large database studies of Type 2 Diabetes show that metformin is related to reducing the risk of dementia, but some studies have different conclusions, and there is few related study in elderly obese patients. The investigators speculate that metformin may improve cognitive dysfunction by improving central insulin resistance in elderly obese patients.

A prospective, randomized controlled single center clinical cohort study will be conducted on 54 elderly obese patients with MCI. One group will receive metformin and lifestyle intervention, while the control group will receive simple lifestyle intervention. All subjects will be followed up for 26 weeks. Medical history collection, physical examination, and laboratory tests will be conducted before and after intervention, and the Montreal Cognitive Assessment Scale will be used for evaluation. Nasal insulin inhalation combined with fMRI will be used to evaluate central insulin resistance status as an objective basis for cognitive function evaluation. The main purpose of the study is to provide more accurate clinical research evidence for the prevention and treatment of MCI in elderly obese patients, in order to reduce the risk of developing dementia and alleviate the burden on families and society.

DETAILED DESCRIPTION:
1. The prevalence of cognitive impairment among elderly obese patients is high, and early intervention for them is of great significance.

   Cognitive impairment refers to the impairment of one or more aspects such as learning and memory, language, executive function, perceptual-motor function, complex attention, and social cognition, often accompanied by mental, behavioral, and personality abnormalities, including mild cognitive impairment (MCI) and dementia. Epidemiological studies have shown that the prevalence of MCI among people aged 60 and above in China is 15.5%, and the affected population reaches 38 million. Numerous studies have confirmed the clear association between obesity and cognitive impairment. The daily life of MCI patients is less interfered by cognitive deficits, but the proportion of their annual progression to dementia can reach 5-10%, which is much higher than the 1-2% incidence rate of the general population. 50% of MCI patients can develop dementia within 5 years and 20-30% of MCI patients can recover normal cognition. Therefore, early detection of MCI in elderly obese patients and timely intervention have important clinical significance and value.
2. Central nervous system insulin resistance plays a role in the pathogenesis of cognitive dysfunction. Functional magnetic resonance imaging(fMRI) can assess cognitive dysfunction by observing central insulin resistance.

   Currently, the mechanisms of cognitive dysfunction in elderly obese patients include the pathological physiological effects of microvascular mechanisms and fat-derived factors. Insulin not only regulates peripheral metabolism but also acts on the central nervous system to regulate cognitive function. All cell types in the brain have an insulin signaling pathway, and studies have shown that brain insulin resistance can damage the plasticity of hippocampal synapses and memory function, thereby leading to cognitive decline. The evaluation of cognitive function is usually conducted using the Montreal Cognitive Assessment Scale(Moca), which includes multiple dimensions such as memory, attention, executive function, and language function, with a maximum score of 30. The score considered for diagnosing MCI is 20-26 (education> 10 years) or 20-25 (education≤ 10 years). However, in practical work, the collection of the scale is affected by many factors. fMRI can show changes in local blood flow and metabolic activities in the brain before brain structure changes, and can deeply understand brain functional changes, which is an important means for early diagnosis of cognitive dysfunction, efficacy monitoring, and mechanism research. By combining fMRI with nasal insulin inhalation, the response of different brain regions to insulin can be observed to assess the degree of central insulin resistance. If there is no neuroimaging or neurophysiological response after nasal insulin inhalation, it indicates the presence of central nervous system insulin resistance. Previous studies have shown that improving the state of central insulin resistance can delay or reverse cognitive decline. Therefore, the central insulin resistance state observed by fMRI can be used as an objective basis for evaluating cognitive function.
3. Metformin may improve cognitive dysfunction by improving the central insulin resistance of elderly obese patients.

Metformin, as the first-line medication for type 2 diabetes, has been widely used. Basic research shows that metformin has the potential to activate the 5'AMP-activated protein kinase (AMPK) pathway, which plays a crucial role in the pathogenesis of dementia. Metformin can improve insulin resistance, reduce neuronal apoptosis, and reduce oxidative stress and inflammatory responses in the brain. Recent studies have shown that the use of metformin is associated with a significant reduction in the risk of dementia in elderly patients with type 2 diabetes. However, these studies were conducted on diabetes patients in large-scale databases, and drawing conclusions by comparing whether metformin was used or not would be affected by many interfering factors. Some earlier studies have shown that long-term use of metformin may even increase the risk of dementia. This may be related to vitamin B12 deficiency, the duration of metformin use, and the course of diabetes. Some small-sample short-term controlled studies have shown that in non-diabetic MCI patients, metformin can penetrate the blood-brain barrier and improve learning, memory, and attention. In conclusion, as a widely used traditional hypoglycemic drug, basic research suggests that metformin can improve central insulin resistance. Clinical studies in diabetes patients suggest a relatively definite possibility of improving cognitive impairment. However, there are currently few studies on the use of metformin to improve cognitive function in elderly overweight or obese patients with MCI.

Therefore, the investigators plan to conduct an intervention using an adequate dose of metformin in elderly overweight or obese patients with MCI, while using patients with simple lifestyle intervention as the control group. The investigators will use fMRI to evaluate the state of central insulin resistance as an objective basis for cognitive function assessment, reducing the limitations of cognitive scales and achieving early detection and intervention of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60 - 75 years old
* Body Mass Index: ≥ 24 kg/m2
* Glycated Hemoglobin < 8.5%
* Moca Scale score: 20-26 points (education> 10 years) or 20-25 points (education≤ 10 years)
* Sign the informed consent form

Exclusion Criteria:

* Any hypoglycemic drugs have been used within 8 weeks prior to enrollment
* Type 1 diabetes
* Unable to undergo central nervous system magnetic resonance examination
* History of alcohol or drug addiction
* Severe gastrointestinal diseases, history of gastrointestinal surgery, severe cardiac or pulmonary dysfunction, malignant tumors and other diseases
* Abnormal liver function (liver enzyme indicators more than 2.5 times the upper limit of the reference range) or abnormal kidney function (estimated glomerular filtration rate< 45 ml/min)
* There are diseases such as cerebral infarction and vascular dementia
* There are conditions judged by the investigator as being unsuitable for enrollment

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
fMRI | 26 weeks
  The insulin sensitivity of the central nervous system in the two groups of subjects before and after treatment is evaluated by nasal inhalation of insulin combined with fMRI.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment Scale (Moca scale) | 26 weeks
  The Moca scale score ranges from 0 to 30. The higher the score, the better the cognitive function. The Moca scale score for mild cognitive impairment ranges from 20 to 26 points (for those with more than 10 years of education) or 20 to 25 points (for those with 10 years or less of education). The investigators compare the scores of the Moca scale before and after the intervention.

OTHER OUTCOMES:
body composition | 26 weeks
  The body composition is measured using Beijing Yueqi BIA. The indicators include weight (kg), skeletal muscle (kg), body fat (kg), body mass index (kg/m2), body fat percentage (%), visceral fat area (cm2), waist-to-hip ratio, and skeletal muscle index (kg/m2). The investigators compare the changes in body composition before and after the intervention.
grip strength | 26 weeks
  The grip strength is evaluated using an electronic grip strength tester. Each hand is tested twice, and the average values are taken. The side with the greater grip strength is selected as the final grip strength. A low grip strength is defined as less than 28 kg for men and less than 18 kg for women. The investigators compare the changes in grip strength before and after the intervention.
glycated hemoglobin | 26 weeks
  The glycated hemoglobin (%) is measured on an empty stomach, and the investigators compare the changes before and after the intervention.
insulin | 26 weeks
  The measurement of insulin (mIU/L) is conducted in the fasting state. The investigators compare the changes before and after the intervention.
C-peptide | 26 weeks
  The measurement of C-peptide (ng/ml) is conducted in the fasting state. The investigators compare the changes before and after the intervention.
blood glucose | 26 weeks
  The measurement of blood glucose (mmol/L) is conducted in the fasting state. The investigators compare the changes before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Tao, Study Director — Huadong Hospital
Locations (1):
- Huadong Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT07395960/Prot_000.pdf
  • Informed Consent Form (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT07395960/ICF_001.pdf